CLINICAL TRIAL: NCT02608619
Title: Pilot Study to Determine Uptake and Biodistribution of 18F-fluorocholine in Histiocytic Disorders by PET Imaging and Biopsy Measurement
Brief Title: Uptake and Biodistribution of 18F-fluorocholine in Histiocytic Disorders by PET Imaging and Biopsy Measurement
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-268
Record Dates: First submitted 2015-11-17; First posted 2015-11-20 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Erdheim-Chester Disease; Langerhans Cell Histiocytosis; Histiocytic Disorders
Keywords: 18F-fluorocholine; Pet imaging; Biopsy; 15-268
MeSH Terms: conditions — Erdheim-Chester Disease; Histiocytosis, Langerhans-Cell | interventions — Biopsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tissue

GROUPS / COHORTS (1):
- PET Imaging: This study will enroll patients who have a clinical diagnosis of a systemic histiocytic disorder, and who are scheduled to undergo confirmatory biopsies of the systemic lesions, that were identified by standard imaging modalities.
  Interventions: Radiation: F-choline PET Scan; Device: FDG-PET; Procedure: biopsy

INTERVENTIONS:
Radiation: F-choline PET Scan
Device: FDG-PET
Procedure: biopsy

SUMMARY:
The main purpose of this study is to discover how 18F-cholineFCH distributes in the body, and see if it can distinguish active histiocytes (tumor) from inflammatory (non- tumor) cells. This tracer has the potential to give the investigators' team more information when trying to identify the tumor cells that are most important to collect with biopsy. In addition, the study will measure levels of 18F-cholineFCH in the biopsy tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Suspected but pathologically unconfirmed diagnosis of Erdheim-Chester disease or Langerhans cell histiocytosis or other histiocytic disorder on the basis of clinical diagnosis, radiologic features, or findings from prior biopsies

Or

* Confirmed diagnosis of Erdheim-Chester disease or Langerhans cell histiocytosis or other histiocytic disorder and requiring additional diagnostic imaging and biopsy to determine mutational status in order to determine therapeutic options.

Exclusion Criteria:

* Inability to undergo or cooperate with PET/CT scan (e.g., claustrophobia)
* Pregnant or nursing female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients for this study will be recruited by physicians from the Departments of Neurology.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
percentage of patients who successfully undergo paired biopsies | 1 year
  The overall histiocyte content will be described in each patient for each paired biopsy: there will be one biopsy that has high 18F-FCH F-choline uptake and one biopsy that has low 18F-FCH F-choline uptake.

CONTACTS AND LOCATIONS:
Overall Officials: Eli Diamond, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memoral Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/